CLINICAL TRIAL: NCT02969590
Title: Regulation of Cervical Mucus Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Leo Han, Instructor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: OHSU IRB 11532
Record Dates: First submitted 2015-05-27; First posted 2016-11-21 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Fertility; Contraception
Keywords: Contraception; Mucus; Cervix; progestin; hormones
MeSH Terms: interventions — Leuprolide; Estrogens; Estradiol; Progesterone; Progestins; Norethindrone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Intervention: Spontaneous Cycle (1 month) (No Intervention): In order to qualify for the intervention phase, subjects needed to demonstrate favorable mucus at ovulation (Insler score of greater than or equal to 10 within 24h of an LH surge) and progesterone level in the luteal phase consistent with ovulation (a single P4 of greater than or equal to 3ng/ ml between days 18-35 of menstrual cycle).
- NET Arm - Norethindrone (4 months) (Active Comparator): This arm will receive Norethindrone (NET) first then experience estradiol withdrawal (E2WD).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
  Interventions: Drug: Leuprolide acetate; Drug: Estrogen and Progesterone Replacement; Drug: Progestin
- E2WD Arm - Estradiol (4 months) (Active Comparator): This arm will experience estradiol withdrawal (E2WD) first and then receive Norethindrone (NET).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches ; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
  Interventions: Drug: Leuprolide acetate; Drug: Estrogen and Progesterone Replacement; Drug: Progestin

INTERVENTIONS:
Drug: Leuprolide acetate — Following this spontaneous cycle, participants received a single intramuscular injection of leuprolide acetate (11.25mg, LupronVR; Abbvie, Chicago, IL), a dose documented to suppress ovarian function for at least 3 months. Ovarian suppression is confirmed with serum E2 less than or equal to 35 pg/ml 21-28 day post-injection.
  Other Names: Lupron
  Arms: E2WD Arm - Estradiol (4 months); NET Arm - Norethindrone (4 months)
Drug: Estrogen and Progesterone Replacement — Replace hormones exogenously to create an artificial cycle
  Other Names: Estradiol (vivelle-dot); Progesterone (prometrium, progestin)
  Arms: E2WD Arm - Estradiol (4 months); NET Arm - Norethindrone (4 months)
Drug: Progestin — Synthetic progestin to assess effects on cervical mucus.
  Other Names: Norethindrone; NET
  Arms: E2WD Arm - Estradiol (4 months); NET Arm - Norethindrone (4 months)

SUMMARY:
The purpose of this study is to help us determine how hormones impact the production of cervical mucus which is a fluid secreted by the opening of the uterus, also called the cervix. During a normal menstrual cycle, cervical mucus changes in response to two hormones that the ovaries make: estrogen and progesterone. Many of the birth control methods women use thicken mucus and make it less likely for sperm to enter the uterus. The goal of this study is to better understand the effects estrogen and progesterone have on the cervical mucus in the body. To do this, the investigators will be using a drug that suppresses natural hormone production for 3 months. Estrogen and progesterone will be artificially replaced to better understand their effects. The investigators will also be studying the effect of a common birth control pill that may work by thickening cervical mucus. Last, the investigators will study some of the cells in the cervix that produce mucus.

DETAILED DESCRIPTION:
This proposed study is to evaluate the temporal changes in human cervical mucus in response to progesterone and progestins as an initial step toward clarifying these relationships. Our hypothesis is that direct effects of progesterone on the endocervix, independent of estrogen withdrawal, cause contraceptive changes to cervical mucus. To study this, a randomized, prospective, crossover study will be conducted by examining cervical mucus changes in a small cohort of women in whom investigators will suppress circulating hormonal levels by administering a GnRH antagonist. Investigators will then artificially replace Estrogen and Progesterone in order to differentiate their effects on clinical and laboratory measurements of mucus quality. The investigators will be looking closely at the immediate changes in mucus when .35 mg of norethindrone, a marketed drug is administered in this experimental setting. Cervical cell samples will also be collected at various time points and perform RT-PCR to determine whether genes for membrane bound progesterone receptor are expressed and regulated by Estrogen and Progesterone.

ELIGIBILITY:
Inclusion Criteria:

* Normal menstrual cycles of 25-35 days in length for at least previous 3 cycles
* 21-40 years of age
* BMI >18, <30
* Serum P4 ≥ 3 ng/ml on single sample collected between days 18-25 of self-reported menstrual cycle
* Flexible schedule allowing morning blood draws on less than 48 hour notice
* In good general health
* Commit to remain on stable diet during study period (no changes to normal dietary habits)
* Commit to using non-hormonal contraceptive methods during study period except those prescribed in the experimental protocol
* No objections to taking study drugs
* No objections to refraining from intercourse the night before any sampling and willing to using condoms during vaginal intercourse.

Exclusion Criteria:

* Oral contraceptive use or other hormone supplement within the preceding 2 months
* Women with current cervical infection
* Evidence of abnormal cervical cytology
* Use of Paragard IUD for contraception
* Long-acting hormonal contraceptive use in the past 12 months (e.g., Depo-Provera®)
* Contraindications to study drugs
* Current or past pregnancy within the previous 6 months or currently trying to conceive
* Desiring to conceive in the next 8 months
* Breastfeeding in the past 2 months
* Diagnosed Diabetes or Metabolic Syndrome
* Current or previous use of cholesterol lowering drugs within the preceding 12 months
* Diagnosed Polycystic Ovary Syndrome
* History of, or self-reported, substance abuse
* Smoker
* Previous infertility treatment excluding male factor issues
* Use of an investigational drug within the past 2 months
* History of excisional or ablative treatment procedure on cervix (ie. LEEP, Cryotherapy, Cold Knife Cone)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03-29 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Han, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Han L, Padua E, Edelman A, Jensen JT. Appraising cervical mucus: a new approach to evaluating contraceptives. Eur J Contracept Reprod Health Care. 2018 Feb;23(1):78-83. doi: 10.1080/13625187.2018.1437134. Epub 2018 Feb 19. PMID 29457758

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to qualify for the intervention phase, subjects needed to demonstrate an ovulatory menstrual cycle during the Screening Period.
Groups:
- Spontaneous Cycle: In order to qualify for the intervention phase, subjects needed to demonstrate favorable mucus at ovulation (Insler score of greater than or equal to 10 within 24h of an LH surge) and progesterone level in the luteal phase consistent with ovulation (a single P4 of greater than or equal to 3ng/ ml between days 18-35 of menstrual cycle).
- NET Arm - Norethindrone, Then Estradiol Withdrawal: This arm will receive Norethindrone (NET) first then experience estradiol withdrawal (E2WD).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
- E2WD Arm - Estradiol Withdrawal, Then Norethindrone: This arm will experience estradiol withdrawal (E2WD) first and then receive Norethindrone (NET).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
Period: Screening Period
Arm/Group | Spontaneous Cycle | NET Arm - Norethindrone, Then Estradiol Withdrawal | E2WD Arm - Estradiol Withdrawal, Then Norethindrone
Started | 5 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Hormones not suppressed post Lupron | 1 | 0 | 0
Period: Treatment Period 1
Arm/Group | Spontaneous Cycle | NET Arm - Norethindrone, Then Estradiol Withdrawal | E2WD Arm - Estradiol Withdrawal, Then Norethindrone
Started | 0 | 2 | 2
Completed | 0 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Spontaneous Cycle | NET Arm - Norethindrone, Then Estradiol Withdrawal | E2WD Arm - Estradiol Withdrawal, Then Norethindrone
Started | 0 | 2 | 2
Completed | 0 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Norethindrone, Then Estradiol Withdrawal: This arm will receive Norethindrone (NET) first then experience estradiol withdrawal (E2WD).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
- Estradiol Withdrawal, Then Norethindrone: This arm will experience estradiol withdrawal (E2WD) first and then receive Norethindrone (NET).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
- Total: Total of all reporting groups
Arm/Group | Norethindrone, Then Estradiol Withdrawal | Estradiol Withdrawal, Then Norethindrone | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Median Cervical Mucus Score - Baseline
Description: Measurement of median cervical mucus scores at baseline. The current clinical standard for appraising cervical mucus is the cervical mucus score (ie. Insler score) that examines mucus based on 5 metrics including volume, spinnbarkeit (stretch), ferning, viscosity and cellularity on a 15-point scale. Per WHO guidelines, scores above 10 are considered "mucus favoring penetration" and scores below 10 are considered to be "unfavorable to penetration."
Time Frame: Baseline
Population: Data from one (1) subject were excluded from analyses because estradiol (E2) levels were consistent with patch noncompliance
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Norethindrone: This arm will receive Norethindrone (NET) first then experience estradiol withdrawal (E2WD).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
- Estradiol: This arm will experience estradiol withdrawal (E2WD) first and then receive Norethindrone (NET).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
Arm/Group | Norethindrone | Estradiol
Number analyzed (Participants) | 3 | 3
score on a scale | 11 [9 to 12] | 13 [12 to 13]

2. Primary Outcome: Sperm Penetration Scores
Description: Measuring sperm penetration scores in different hormonal conditions
Time Frame: Approximately one year
Population: Outcome not analyzed.
Arm/Group | Norethindrone | Estradiol
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in PGRMC1 During Menstrual Cycle
Description: Measuring the mean transcript change of membrane bound progestin receptors (PGRMC1) from follicular phase to ovulation to luteal phase of spontaneous menstrual cycle.
  Total RNA (ribonucleic acid) was isolated from endocervical cell samples and analyzed for expression of PGRMC1 using real-time PCR (polymerase chain reaction) relative to levels of ribosomal (S10) RNA. An endocervical brush will be inserted into the os and then immediately rinsed into a special RNA preserving reagent. After total RNA is isolated and purified, it will be reverse transcribed into cDNA using primers.
  Ratio of PGRMC1 to 18s RNA
  Gene expression of membrane bound progesterone receptors in endocervical cells
Time Frame: 1 month
Population: PGRMC1 data was analyzed for the 4 subjects who demonstrate ovarian suppression following leuprolide injection and continued to intervention phase of the study. Outcome was only evaluated during spontaneous menstrual cycle (1 month).
  One participant corresponds to one cycle.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Spontaneous Cycle: In order to qualify for the intervention phase, subjects needed to demonstrate favorable mucus at ovulation (Insler score of greater than or equal to 10 within 24h of an LH surge) and progesterone level in the luteal phase consistent with ovulation (a single P4 of greater than or equal to 3ng/ ml between days 18-35 of menstrual cycle).
  Prior to the intervention cycle, each subject was observed over the normal natural cycle during which time we collected menstrual data including serum sex-steroid levels, mucus and cytology brushings for PGRMC1 analysis.
Arm/Group | Spontaneous Cycle | Norethindrone | Estradiol
Number analyzed (Participants) | 4 | 0 | 0
ratio
  Follicular Phase | 1.2 (0.38) |  |
  Ovulation Phase | 4.0 (2.4) |  |
  Luteal Phase | 1.02 (0.73) |  |

4. Primary Outcome: Median Cervical Mucus Score - 2 Hour
Description: Measurement of median cervical mucus scores 2 hours following norethindrone administration. The current clinical standard for appraising cervical mucus is the cervical mucus score (ie. Insler score) that examines mucus based on 5 metrics including volume, spinnbarkeit (stretch), ferning, viscosity and cellularity on a 15-point scale. Per WHO guidelines, scores above 10 are considered "mucus favoring penetration" and scores below 10 are considered to be "unfavorable to penetration."
Time Frame: 2 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Norethindrone | Estradiol
Number analyzed (Participants) | 3 | 3
score on a scale | 8.5 [4 to 9] | 10.5 [10 to 12]

5. Primary Outcome: Median Cervical Mucus Score - 6 Hour
Description: Measurement of median cervical mucus scores 6 hours following norethindrone administration. The current clinical standard for appraising cervical mucus is the cervical mucus score (ie. Insler score) that examines mucus based on 5 metrics including volume, spinnbarkeit (stretch), ferning, viscosity and cellularity on a 15-point scale. Per WHO guidelines, scores above 10 are considered "mucus favoring penetration" and scores below 10 are considered to be "unfavorable to penetration."
Time Frame: 6 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Norethindrone | Estradiol
Number analyzed (Participants) | 3 | 3
score on a scale | 6.5 [6 to 8] | 8.5 [8 to 9]

6. Primary Outcome: Median Cervical Mucus Score - 24 Hour
Description: Measurement of median cervical mucus scores 24 hours following norethindrone administration. The current clinical standard for appraising cervical mucus is the cervical mucus score (ie. Insler score) that examines mucus based on 5 metrics including volume, spinnbarkeit (stretch), ferning, viscosity and cellularity on a 15-point scale. Per WHO guidelines, scores above 10 are considered "mucus favoring penetration" and scores below 10 are considered to be "unfavorable to penetration."
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Norethindrone | Estradiol
Number analyzed (Participants) | 3 | 3
score on a scale | 8 [7 to 8] | 10.5 [8 to 11]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Crossover study. One participant corresponds to one cycle.
Groups:
- Spontaneous Cycle: Adverse Events experienced by subjects during Spontaneous Cycle.
  In order to qualify for the intervention phase, subjects needed to demonstrate favorable mucus at ovulation (Insler score of greater than or equal to 10 within 24h of an LH surge) and progesterone level in the luteal phase consistent with ovulation (a single P4 of greater than or equal to 3ng/ ml between days 18-35 of menstrual cycle).
- Norethindrone (NET): Adverse Events experienced by subjects for the Norethindrone intervention (while in the Norethindrone (NET) arm of study).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
- Estradiol (E2): Adverse Events experienced by subjects for the Estradiol (E2) intervention (while in the estradiol (E2) arm of study).
  On the day prior to each admission, we instructed subjects to apply three fresh estradiol (E2) patches (0.3mg/day) to achieve mid-cycle level E2 effects.
  On the day of the first and third admission, subjects were randomized to the experimental condition, either: (1) oral progestin administration (e.g., a single dose of 0.35mg norethindrone) with continuation of the E2 patches; or (2) estradiol withdrawal (e.g., removal of the patches). Subject then received the converse intervention for admissions two and four.
  Subjects resumed treatment with the 0.1mg E2 patch until their next scheduled inpatient assessment. We required a minimum of five days at this level before repeating the dose escalation and the next evaluation.
Arm/Group | Spontaneous Cycle | Norethindrone (NET) | Estradiol (E2)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT02969590/Prot_SAP_000.pdf